CLINICAL TRIAL: NCT07064707
Title: Clinical Study to Evaluate Safety and Efficacy of Rupatadine in Patients With Ulcerative Colitis.
Brief Title: Rupatadine in Patients With Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Prof. Dr. Ahmed Ibrahim Mohammed El Mallah, faculty of pharmacy, Alexandria University. (Unknown); Assoc. Prof. Dr. Noha Alaa Eldin Hassan Hamdy, Faculty of pharmacy, Alexandria University. (Unknown); Assoc. Prof. Dr. Ibrahim Fathi Amer, Faculty of Medecine, Kafr Elsheikh University. (Unknown)
Responsible Party: Principal Investigator, Reham ELshafeiy, Associate lecturer of clinical pharmacy, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5555
Record Dates: First submitted 2025-07-06; First posted 2025-07-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; rupatadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): control group (Mesalamine group) who will receive 1 g mesalamine three times daily for 3 months.
  Interventions: Drug: Mesalamine
- Rupatadine (Active Comparator): (Rupatadine group) will receive 1 g mesalamine three times daily plus 20 mg rupatadine once daily for 3 months.
  Interventions: Drug: Mesalamine; Drug: Rupatadine

INTERVENTIONS:
Drug: Mesalamine — Mesalamine or 5-amino salicylic acid (5-ASA), plays a crucial role in the treatment of ulcerative colitis (UC). It is the first-line therapy for mild to moderate cases of UC and is considered a cornerstone in its management.
Drug: Rupatadine — Rupatadine, a dual histamine H1 receptor and platelet-activating factor (PAF) receptor antagonist, has shown promising anti-inflammatory effects beyond its conventional use in allergic conditions
  Arms: Rupatadine

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory condition that primarily targets the large intestine. Although substantial progress has been made in treatment modalities-especially with the development of immunomodulatory drugs and biologic therapies-managing UC continues to present significant challenges. At present, there is no definitive cure, and current treatment strategies are largely focused on controlling inflammation, relieving symptoms, and halting disease progression

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Both male and female will be included
* Mild and moderate UC patients are already diagnosed and confirmed by endoscope and histopathology.

Exclusion criteria:

* Breast feeding or pregnancy.
* Colorectal cancer patients.
* Patients with severe UC.
* Patients taking rectal or systemic steroids.
* Patients taking immunosuppressives or biological therapies.
* Addiction to alcohol and / or drugs.
* Known allergy to the studied medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
change in partial mayo score | 3 months
  The Partial Mayo Score (PMS) index will be utilized to ascertain the degree of disease severity. One non-invasive clinical measure for determining the severity of UC is the PMS. The composite score is derived from three subcategories: stool frequency, rectal bleeding, and physician's general assessment. The total score falls between 0 and 9

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt